CLINICAL TRIAL: NCT00133302
Title: Randomized Phase III Study of Standard CHOP (S-CHOP) Versus Biweekly CHOP (Bi-CHOP) in Aggressive Non-Hodgkin's Lymphoma (JCOG9809)
Brief Title: Study of Standard CHOP Versus Biweekly CHOP in Aggressive Non-Hodgkin's Lymphoma (JCOG9809)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9809; C000000036
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2006-08

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's lymphoma; intermediate-grade lymphoma; high-grade lymphoma; CHOP protocol; granulocyte-colony stimulating factor
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Drug: Standard CHOP
Drug: Bi-CHOP (dose intensified CHOP)

SUMMARY:
The purpose of this trial is to investigate the clinical benefit of the dose intensified regimen, Bi-CHOP in comparison to standard CHOP for advanced intermediate or high grade non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
The purpose of JCOG9809 was to determine whether treatment results of aggressive NHL could be improved by shortening intervals of CHOP chemotherapy with the prophylactic use of G-CSF. The primary endpoint was Progression Free Survival (PFS), and the planned accrual was 450. Until December, 2002, 323 patients with advanced aggressive NHL were randomized to standard CHOP arm (CHOP x 8, every three weeks) and biweekly CHOP arm (CHOP x 8, every two weeks).

ELIGIBILITY:
Inclusion Criteria:

* Intermediate- or high-grade non-Hodgkin's lymphoma, excluding cutaneous t-cell lymphoma (CTCL), adult T-cell leukemia-lymphoma (ATL) and T-cell lymphoblastic lymphoma (T-LbL) (Working Formulation)
* Ann Arbor stage: II, III, IV
* No prior chemotherapy or radiotherapy
* Age: 15 to 69
* Performance status (PS): 0, 1, 2
* WBC >= 3,000 /mm3, ANC >= 1,200 /mm3, Platelet >= 75,000 /mm3
* GOT/GPT <= 5 x Normal Upper Limit, T-Bil <= 2.0 mg/dL
* Creatinine <= 2.0 mg/dL
* Normal ECG, Ejection Fraction >= 50%
* PaO2 >= 65 mmHg
* Written informed consent

Exclusion Criteria:

* Uncontrollable diabetes mellitus
* Severe complication (infection, heart failure, renal failure, liver failure, etc)
* Anamnesis of heart disease
* Acute or chronic hepatitis, liver cirrhosis and portal hypertension
* Synchronous or metachronous malignancy
* Severe pulmonary dysfunction
* Central nervous system (CNS) invasion
* HIV positive
* Hepatitis B surface antigen (HBs-Ag) positive
* Hepatitis C virus antibody (HCV-Ab) positive

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 1999-02; Study Completion 2005-02

PRIMARY OUTCOMES:
Progression free survival

SECONDARY OUTCOMES:
Overall survival
Complete remission rate
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Tomomitsu Hotta, MD, PhD, Study Chair — Tokai University
Locations (1):
- Tokai University, Isehara, Kanagawa, Japan

REFERENCES:
- [Derived] Ohmachi K, Tobinai K, Kobayashi Y, Itoh K, Nakata M, Shibata T, Morishima Y, Ogura M, Suzuki T, Ueda R, Aikawa K, Nakamura S, Fukuda H, Shimoyama M, Hotta T; members of the Lymphoma Study Group of the Japan Clinical Oncology Group (JCOG-LSG). Phase III trial of CHOP-21 versus CHOP-14 for aggressive non-Hodgkin's lymphoma: final results of the Japan Clinical Oncology Group Study, JCOG 9809. Ann Oncol. 2011 Jun;22(6):1382-1391. doi: 10.1093/annonc/mdq619. Epub 2010 Dec 31. PMID 21196441
- See also: Related Info — http://www.jcog.jp/